CLINICAL TRIAL: NCT01482338
Title: A Comparative Efficacy of Low-dose Combine Oral Contraceptives Containing Desogestrel 150 mg and Drospirenone 3 mg on Premenstrual Symptoms
Brief Title: Premenstrual Symptoms Treatment Comparing Between Oral Contraceptives Containing Desogestrel and Drospirenone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jirath Wichianpitaya,MD., Mr, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMS 068/54
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; Low-dose combine contraceptives pills; COC
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Desogestrel; ethinyl estradiol-desogestrel combination; drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSG (Experimental): The low-dose oral contraceptive pill which one consists of 20 microgram ethinyl estradiol and 150 mg desogestrel were taken orally by participants every day beginning Day1 to Day 3 of the first menstrual cycle until complete 24 days and continued with free-hormone pills for 4 days. The next cycle has to continue in the same way until complete 6 cycles.
  Interventions: Drug: EE 20 microgram with desogestrel 150 mg
- DRSP (Active Comparator): The other low-dose oral contraceptive pill which consists of 20 microgram ethinyl estradiol and 3 mg drospirenone were taken orally by participants every day beginning Day1 to Day 3 of the first menstrual cycle until complete 24 days and continued with free-hormone pills for 4 days. The next cycle has to continue in the same way until complete 6 cycles.
  Interventions: Drug: EE 20 microgram with drospirenone 3 mg

INTERVENTIONS:
Drug: EE 20 microgram with desogestrel 150 mg — Comparison of 2 different low-dose oral contraceptive pill which one consists of 20 microgram ethinyl estradiol and 150 mg desogestrel and the other consists of 20 microgram ethinyl estradiol and 3 mg drospirenone. Both were taken orally by participants every day beginning Day1 to Day 3 of the first menstrual cycle until complete 24 days and continued with free-hormone pills for 4 days. The next cycle has to continue in the same way until complete 6 cycles.
  Other Names: Mercilon
  Arms: DSG
Drug: EE 20 microgram with drospirenone 3 mg — Comparison of 2 different low-dose oral contraceptive pill which one consists of 20 microgram ethinyl estradiol and 150 mg desogestrel and the other consists of 20 microgram ethinyl estradiol and 3 mg drospirenone. Both were taken orally by participants every day beginning Day1 to Day 3 of the first menstrual cycle until complete 24 days and continued with free-hormone pills for 4 days. The next cycle has to continue in the same way until complete 6 cycles.
  Other Names: Yaz
  Arms: DRSP

SUMMARY:
The purpose of this study is to determine whether low-dose combine oral contraceptives (COC) containing desogestrel 150 mg and drospirenone 3 mg are effective in the treatment of Premenstrual symptoms.

DETAILED DESCRIPTION:
Premenstrual syndrome is commonly reported 20-90 percent in reproductive-aged women. Only a small percentage of women (2 to 5%) have significant premenstrual symptoms defined as Premenstrual dysphoric disorder (PMDD). The exact symptoms and their intensity vary from woman to woman and even from cycle to cycle.While exact causes of PMS are not fully understood,current thinking suspects that fluctuation of endogenous sex hormones are relevant. The standard 21/7 design may induce menstrual-related symptoms including headache, mood swings, abdominal cramping, bloating, and breast tenderness that increase during the last week of active pills extending along the 7-day hormone free interval(HFI). The decline in endogenous estradiol levels during HFI may be responsible for the estrogen-withdrawal symptoms. While a new COC with drospirenone introduced in 24/4 design has been shown in clinical trials to significantly improve the symptoms of PMS, there has been questioned about efficacy of the other kind of COC which has optimal properties, for example, good-control cycles extend to the similar 24/4 regimen.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35years
* Regular menses, I:21-35 days
* Willingness to take COC for 6 months
* No history of COC in last 6 months
* No history of injected contraception in last 6 months
* History of implant contraception need to have regular menses 3 cycles
* History of miscarriage need to have regular menses 3 cycles

Exclusion Criteria:

* Pregnant or suspected pregnant
* Breast feeding
* Smoking
* Contraindication of WHO 2,3 and 4
* PMDD

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Women's Health Assessment Questionnaire (WHAQ)score | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jirath Wichianpitaya, M.D., Principal Investigator — Chulalongkorn University; Surasak Taneepanichskul, M.D., Study Chair — Chulalongkorn University
Locations (1):
- Family Unit, King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Sveindottir H, Backstrom T. Prevalence of menstrual cycle symptom cyclicity and premenstrual dysphoric disorder in a random sample of women using and not using oral contraceptives. Acta Obstet Gynecol Scand. 2000 May;79(5):405-13. doi: 10.1080/j.1600-0412.2000.079005405.x. PMID 10830769
- [Background] Kurshan N, Neill Epperson C. Oral contraceptives and mood in women with and without premenstrual dysphoria: a theoretical model. Arch Womens Ment Health. 2006 Jan;9(1):1-14. doi: 10.1007/s00737-005-0102-z. Epub 2005 Oct 5. PMID 16206030
- [Background] Winer SA, Rapkin AJ. Premenstrual disorders: prevalence, etiology and impact. J Reprod Med. 2006 Apr;51(4 Suppl):339-47. PMID 16734317
- [Background] Paoletti AM, Lello S, Fratta S, Orru M, Ranuzzi F, Sogliano C, Concas A, Biggio G, Melis GB. Psychological effect of the oral contraceptive formulation containing 3 mg of drospirenone plus 30 microg of ethinyl estradiol. Fertil Steril. 2004 Mar;81(3):645-51. doi: 10.1016/j.fertnstert.2003.08.030. PMID 15037415
- [Background] New PMS guidelines released. Recommendations focus on diagnosis and treatment. AWHONN Lifelines. 2000 Jun-Jul;4(3):61-2. doi: 10.1111/j.1552-6356.2000.tb01435.x. PMID 11249391
- [Background] Moos RH. Typology of menstrual cycle symptoms. Am J Obstet Gynecol. 1969 Feb 1;103(3):390-402. doi: 10.1016/0002-9378(69)90499-2. No abstract available. PMID 5812581
- [Background] Spona J, Elstein M, Feichtinger W, Sullivan H, Ludicke F, Muller U, Dusterberg B. Shorter pill-free interval in combined oral contraceptives decreases follicular development. Contraception. 1996 Aug;54(2):71-7. doi: 10.1016/0010-7824(96)00137-0. PMID 8842582
- [Background] Tuckwell P. Schooling the subnormal child. The Massachusetts System. Nurs Mirror Midwives J. 1975 Sep 18;141(12):73-4. No abstract available. PMID 1042815
- [Background] Pearlstein TB, Bachmann GA, Zacur HA, Yonkers KA. Treatment of premenstrual dysphoric disorder with a new drospirenone-containing oral contraceptive formulation. Contraception. 2005 Dec;72(6):414-21. doi: 10.1016/j.contraception.2005.08.021. Epub 2005 Nov 2. PMID 16307962
- [Background] Winkler UH, Ferguson H, Mulders JA. Cycle control, quality of life and acne with two low-dose oral contraceptives containing 20 microg ethinylestradiol. Contraception. 2004 Jun;69(6):469-76. doi: 10.1016/j.contraception.2003.12.017. PMID 15157791
- [Background] Sulak PJ, Carl J, Gopalakrishnan I, Coffee A, Kuehl TJ. Outcomes of extended oral contraceptive regimens with a shortened hormone-free interval to manage breakthrough bleeding. Contraception. 2004 Oct;70(4):281-7. doi: 10.1016/j.contraception.2004.04.007. PMID 15451331
- [Background] Lopez LM, Kaptein AA, Helmerhorst FM. Oral contraceptives containing drospirenone for premenstrual syndrome. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006586. doi: 10.1002/14651858.CD006586.pub3. PMID 19370644
- [Background] Sulak PJ, Scow RD, Preece C, Riggs MW, Kuehl TJ. Hormone withdrawal symptoms in oral contraceptive users. Obstet Gynecol. 2000 Feb;95(2):261-6. doi: 10.1016/s0029-7844(99)00524-4. PMID 10674591